CLINICAL TRIAL: NCT02981524
Title: A Phase 2 Study of GVAX Colon Vaccine (With Cyclophosphamide) and Pembrolizumab in Patients With Mismatch Repair-Proficient (MMR-p) Advanced Colorectal Cancer
Brief Title: Study of GVAX (With CY) and Pembrolizumab in MMR-p Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J16154; IRB00114053 (Other: JHMIRB); MISP53919 (Other: Merck and Company)
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases; Colonic Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases; Colonic Diseases | interventions — Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CY/GVAX with Pembrolizumab (Experimental): During each 21 day cycles, Cyclophosphamide (CY) is administered on Day 1 at 200 mg/m2 followed by Pembrolizumab at 200mg, the colon cancer vaccine (GVAX) is administered on Day 2 at 5E8 colon cancer cells + 5E7 GM-CSF secreting cells for the first 4 cycles of treatment. After cycle 4, cyclophosphamide and GVAX will be administered with every 4th cycle.
  Interventions: Drug: CY; Biological: GVAX; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CY — CY is administered intravenously at 200 mg/m2
  Other Names: Cyclophosphamide, Cytoxan
Biological: GVAX — GVAX is administered intradermally at 5E8 colon cancer cells + 5E7 GM-CSF secreting
  Other Names: Colon cancer vaccine
Drug: Pembrolizumab — Pembrolizumab is administered intravenously at 200 mg
  Other Names: KEYTRUDA, MK-3475

SUMMARY:
This study will be looking at the objective response rate (ORR) as measured by RECIST in in patients with mismatch repair-proficient (MMR-p), advanced colorectal cancer that treated with CY/GVAX in combination with Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Documented mismatch repair-proficient cancer of colorectum, who have received at least two prior lines of therapy for metastatic disease
2. Measurable disease by RECIST v1.1
3. Age >18 years
4. ECOG Performance Status of 0 to 1
5. Estimated life expectancy of greater than 3 months.
6. Adequate organ function as defined by study-specified laboratory tests
7. Must use acceptable form of birth control through the study and for 120 days after final dose of study drug
8. Signed informed consent form
9. Willing and able to comply with study procedures

Exclusion Criteria:

1. Has a known additional malignancy that is progressing or requires active treatment.
2. Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Has known malignant small bowel obstruction within the last 6 months.
4. Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions.
5. Systemically active steroid use.
6. Has an active infection requiring systemic therapy.
7. Has a known history of active TB (Bacillus Tuberculosis).
8. Infection with HIV or hepatitis B or C.
9. Has history of (non-infectious) pneumonitis that required steroids.
10. Must not require supplemental oxygen or have a pulse oximetry < 92% on room air.
11. Conditions, including therapy, laboratory abnormalities, psychiatric or substance abuse disorders, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures.
12. Pregnant or lactating.
13. Another investigational product within 28 days prior to receiving study drug.
14. Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug.
15. Chemotherapy, radiation, hormonal, or biological cancer therapy within 28 days prior to receiving study drug.
16. Has received a live vaccine within 30 days of planned start of study therapy.
17. Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.).
18. Patients receiving growth factors including, but not limited to, granulocyte-colony stimulating factor (G-CSF), GM-CSF, erythropoietin, within 14 days of study drug administration.
19. Hypersensitivity to pembrolizumab or any of its excipients.
20. Patient has a known or suspected hypersensitivity to GM-CSF, hetastarch, corn, dimethyl sulfoxide, fetal bovine serum, trypsin (porcine origin), yeast or any other component of GVAX vaccine.
21. Presence of any tissue or organ allograft and history of allogeneic hematopoietic stem cell transplant.
22. Unwilling or unable to comply with study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yarchoan M, Huang CY, Zhu Q, Ferguson AK, Durham JN, Anders RA, Thompson ED, Rozich NS, Thomas DL 2nd, Nauroth JM, Rodriguez C, Osipov A, De Jesus-Acosta A, Le DT, Murphy AG, Laheru D, Donehower RC, Jaffee EM, Zheng L, Azad NS. A phase 2 study of GVAX colon vaccine with cyclophosphamide and pembrolizumab in patients with mismatch repair proficient advanced colorectal cancer. Cancer Med. 2020 Feb;9(4):1485-1494. doi: 10.1002/cam4.2763. Epub 2019 Dec 26. PMID 31876399

RESULTS

PARTICIPANT FLOW:
Groups:
- CY/GVAX With Pembrolizumab: During each 21 day cycles, Cyclophosphamide (CY) is administered on Day 1 at 200 mg/m2 followed by Pembrolizumab at 200mg, the colon cancer vaccine (GVAX) is administered on Day 2 at 5E8 colon cancer cells + 5E7 GM-CSF secreting cells.
  CY: CY is administered intravenously at 200 mg/m2
  GVAX: GVAX is administered intradermally at 5E8 colon cancer cells + 5E7 GM-CSF secreting
  Pembrolizumab: Pembrolizumab is administered intravenously at 200 mg
Period: Overall Study
Arm/Group | CY/GVAX With Pembrolizumab
Started | 17
Completed | 0
Not Completed | 17
Not completed — Progressive Disease | 14
Not completed — Death (unrelated) | 1
Not completed — Treatment Related Toxicity | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | CY/GVAX With Pembrolizumab
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased
  Participants
    ECOG 0 | 6
    ECOG 1 | 11
Baseline Carcinoembryonic Antigen (CEA) [Median (Inter-Quartile Range); unit: ng/ml] | 84.8 [51.4 to 333.9]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: up to 1 year
Population: Data to assess objective response was only collected from 14/17 participants. The remaining 3 patients were withdrawn from study therapy for early clinical progression and were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CY/GVAX With Pembrolizumab
Number analyzed (Participants) | 14
Participants | 0

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of participants who experience treatment related adverse events ≥ grade 3 as defined by CTCAE 4.0.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CY/GVAX With Pembrolizumab
Number analyzed (Participants) | 17
Participants | 6

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free Survival (PFS) is defined as the number of days from cycle 1, day 1 of immunotherapy until first documented local progression or death due to any cause. PD is >20% increase in sum of diameters of target lesions as assessed using RECIST (version 1.1).
Time Frame: up to 1 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CY/GVAX With Pembrolizumab
Number analyzed (Participants) | 17
days | 82 [48 to 97]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the number of days from start of study treatment to time of death. Individuals will be censored at the date of the last study visit if no event occurs. The estimation method used was Kaplan-Meier.
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CY/GVAX With Pembrolizumab
Number analyzed (Participants) | 17
days | 213 [179 to 441]

5. Secondary Outcome: Duration of Response (DOR)
Description: Number of weeks from the start date of PR or CR (whichever response is recorded first) and subsequently confirmed to the first date that recurrent or progressive disease or death is documented. Per RECIST 1.1, CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions.
Time Frame: 1 year
Population: There were no patients that had a CR or PR. Therefore, data could not be collected to assess this outcome measure.
Arm/Group | CY/GVAX With Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse reporting collection was conducted by regular investigator assessment and laboratory measurements.
Arm/Group | CY/GVAX With Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 14/17
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CY/GVAX With Pembrolizumab (N=17)
Eye disorders-Corneal transplant rejection (Eye disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Death, Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms, progression (Brain metastases) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CY/GVAX With Pembrolizumab (N=17)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hemolytic anemia (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4)
Blurred vision (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema-limbs (General disorders) | 3 (3) — and administration site conditions
Fatigue (General disorders) | 4 (4) — and administration site conditions
Fever (General disorders) | 2 (2) — and administration site conditions
Flu-like symptoms (General disorders) | 5 (5) — and administration site conditions
Pain (General disorders) | 10 (10) — and administration site conditions
Fall (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
AST increased (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary pain (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Erectile dysfuntion (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bruising, vaccine site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis, nightsweats (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, vaccine site reaction (Skin and subcutaneous tissue disorders) | 15 (15)
Induration, vaccine site reaction (Skin and subcutaneous tissue disorders) | 16 (16)
Pain, vaccine site reaction (Skin and subcutaneous tissue disorders) | 3 (3)
Macular papular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis, vaccine site reaction (Skin and subcutaneous tissue disorders) | 15 (15)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Warmth, vaccine site reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Hot Flashes (Vascular disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT02981524/Prot_SAP_000.pdf